CLINICAL TRIAL: NCT00026936
Title: A Pilot Study to Investigate the Clinical Utility of the Peregrine Monte Carlo Dose Calculation System for Radiation Therapy Treatment Planning
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990116; 99-C-0116
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Neoplasm
Keywords: External Beam Radiotherapy; TCP; DVH; NTCP; 3-D Programming
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: Radiotherapy

SUMMARY:
The utility of PEREGRINE Monte Carlo calculations for radiation treatment planning in a clinical setting will be assessed by comparing results with other fully three-dimensional programs. ROB will investigate PEREGRINE for clinical use at NCI in collaboration with Lawrence Livermore National Laboratory (LLNL).

DETAILED DESCRIPTION:
The utility of PEREGRINE Monte Carlo calculations for radiation treatment planning in a clinical setting will be assessed by comparing results with other fully three-dimensional programs. ROB will investigate PEREGRINE for clinical use at NCI.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with documented malignancy requiring standard radiotherapy OR patients with a benign condition for whom radiotherapy is indicated.

EXCLUSION CRITERIA:

Documented connective tissue disease or Ataxia Telangiectasia.

Cognitively impaired patients who cannot give informed consent.

Other medical conditions deemed by the PI to make the patient ineligible.

Patients requiring emergent radiotherapy.

Patients who are not able to undergo a CT scan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140
Dates: Start 1999-05; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Perez CA, Purdy JA, Harms W, Gerber R, Graham MV, Matthews JW, Bosch W, Drzymala R, Emami B, Fox S, et al. Three-dimensional treatment planning and conformal radiation therapy: preliminary evaluation. Radiother Oncol. 1995 Jul;36(1):32-43. doi: 10.1016/0167-8140(95)01566-y. PMID 8525023
- [Background] Lawrence TS, Ten Haken RK, Kessler ML, Robertson JM, Lyman JT, Lavigne ML, Brown MB, DuRoss DJ, Andrews JC, Ensminger WD, et al. The use of 3-D dose volume analysis to predict radiation hepatitis. Int J Radiat Oncol Biol Phys. 1992;23(4):781-8. doi: 10.1016/0360-3016(92)90651-w. PMID 1618671
- [Background] Yorke ED, Kutcher GJ, Jackson A, Ling CC. Probability of radiation-induced complications in normal tissues with parallel architecture under conditions of uniform whole or partial organ irradiation. Radiother Oncol. 1993 Mar;26(3):226-37. doi: 10.1016/0167-8140(93)90264-9. PMID 8316652